CLINICAL TRIAL: NCT03849040
Title: Development and Validation of a Computer-aided Algorithm Using Artificial Intelligence and Deep Neural Networks for the Segmentation of Ultrasonographic Features of Lymph Nodes During Endobronchial Ultrasound
Brief Title: The Use of Artificial Intelligence to Predict Cancerous Lymph Nodes for Lung Cancer Staging During Ultrasound Imaging
Status: Completed | Type: Observational
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Wael Hanna, Dr. Waël Hanna, MDCM, MBA, FRCSC, St. Joseph's Healthcare Hamilton
Other Study IDs: StJoes EBUS AI (5636)
Record Dates: First submitted 2019-02-19; First posted 2019-02-21 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Lung Diseases; Lung Neoplasm
Keywords: endobronchial ultrasound; ultrasonographic features; artificial intelligence; deep neural network; segmentation
MeSH Terms: conditions — Lung Diseases; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Endobronchial Ultrasound — All patients will undergo EBUS-TBNA as per routine care, except for the one difference where the procedures will be video-recorded so that they can be used for computer analysis at a later time. Static images will be obtained from EBUS videos in order to perform segmentation. Segmentation will be conducted by both an experienced endoscopist and NeuralSeg.
  Other Names: NeuralSeg

SUMMARY:
This study aims to determine if a deep neural artificial intelligence (AI) network (NeuralSeg) can learn how to assign the Canada Lymph Node Score to lymph nodes examined by endobronchial ultrasound transbronchial needle aspiration(EBUS-TBNA), using the technique of segmentation. Images will be created from 300 lymph nodes videos from a prospective library and will be used as a derivation set to develop the algorithm. An additional100 lymph node images will be prospectively collected to validate if NeuralSeg can correctly apply the score.

ELIGIBILITY:
Inclusion Criteria:

* must be diagnosed with confirmed or suspected lung cancer and be undergoing EBUS diagnosis/staging

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Phase A does not require patient enrollment. Phase B will require prospective enrollment of patients to obtain the validation set of new lymph node videos. All patients who are scheduled to undergo an EBUS-TBNA procedure for mediastinal staging of NSCLC at St. Joseph's Healthcare Hamilton will be eligible to enroll in this study. There are no exclusion criteria. All patients will undergo EBUS-TBNA as per routine care, except for the one difference where the procedures will be video-recorded so that they can be used for computer analysis at a later time.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2019-09-23 (Actual); Study Completion 2019-11-20 (Actual)

PRIMARY OUTCOMES:
Development of computer algorithm to identify lymph node ultrasonographic features | From retrospective data collection to algorithm development (1 month)
  Objective: to determine whether a deep neural AI network (NeuralSeg) can learn how to assign the Canada Lymph Node Score to lymph nodes examined by EBUS, using the technique of segmentation on an existing (derivation) set of lymph node videos
Validation of computer algorithm to identify lymph node ultrasonographic features | From prospective data collection to algorithm validation (6 months)
  Objective: to determine whether NeuralSeg can correctly apply the Canada Lymph Node Score to a new (validation) set of lymph node videos that it has never seen before

SECONDARY OUTCOMES:
Accuracy and reliability of the segmentation performed by NeuralSeg | From segmentation performed by surgeon to segmentation performed by NeuralSeg (1 month)
  Objective: to compare the accuracy and reliability of the segmentation performed by NeuralSeg to the segmentation performed by an experienced endoscopic surgeon using DICE-SORENSEN coefficients.
NeuralSeg prediction of lymph node malignancy | From NeuralSeg algorithm used on EBUS imaging to biopsy report (estimated up to 2-3 months)
  Objective: to determine whether NeuralSeg can accurately predict malignancy in lymph node when compared to biopsy results of the lymph node that was examined.

CONTACTS AND LOCATIONS:
Overall Officials: Wael C Hanna, Principal Investigator — St. Josephs Healthcare Hamilton
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American College of Chest Physicians; Health and Science Policy Committee. Diagnosis and management of lung cancer: ACCP evidence-based guidelines. American College of Chest Physicians. Chest. 2003 Jan;123(1 Suppl):D-G, 1S-337S. No abstract available. PMID 12527560
- [Background] Hanna WC, Yasufuku K. Bronchoscopic staging of lung cancer. Ther Adv Respir Dis. 2013 Apr;7(2):111-8. doi: 10.1177/1753465812468041. Epub 2012 Dec 20. PMID 23258501
- [Background] Hylton DA, Turner J, Shargall Y, Finley C, Agzarian J, Yasufuku K, Fahim C, Hanna WC. Ultrasonographic characteristics of lymph nodes as predictors of malignancy during endobronchial ultrasound (EBUS): A systematic review. Lung Cancer. 2018 Dec;126:97-105. doi: 10.1016/j.lungcan.2018.10.020. Epub 2018 Oct 30. PMID 30527199
- [Background] Topol EJ. High-performance medicine: the convergence of human and artificial intelligence. Nat Med. 2019 Jan;25(1):44-56. doi: 10.1038/s41591-018-0300-7. Epub 2019 Jan 7. PMID 30617339
- [Background] El-Sherief AH, Lau CT, Wu CC, Drake RL, Abbott GF, Rice TW. International association for the study of lung cancer (IASLC) lymph node map: radiologic review with CT illustration. Radiographics. 2014 Oct;34(6):1680-91. doi: 10.1148/rg.346130097. PMID 25310423